CLINICAL TRIAL: NCT01886131
Title: Subthalamic Nuclei (STN) Local Field Potentials to Investigate Motor Control During REM Sleep Behaviour Disorder (TCSP) Secondary to Idiopathic Parkinsons Disease (PD)
Brief Title: Motor Control During Rapid Eye Movement (REM) Sleep Behaviour Disorder
Acronym: RevesParkNST
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Grenoble Institut des Neurosciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 12 388 02; AOL2012 (Other: Toulouse University Hospital)
Record Dates: First submitted 2013-06-20; First posted 2013-06-25 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Parkinson Disease
Keywords: REM behaviour disorder; Subthalamic nucleus; Local field potential; Motor control
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Synchronised video-polysomnography (Experimental)
  Interventions: Other: Synchronised video-polysomnography

INTERVENTIONS:
Other: Synchronised video-polysomnography — We will record the electrical activity of the STN (local field potentials) during the 2 consecutive nights following the implantation of the electrodes in the STN for DBS. In this period, the deep brain stimulator will not yet be connected to the intracranial electrodes.
  The intracranial EEG signal from the STN will be synchronised with the scalp EEG and other video-polysomnographic parameters.
  The STN recordings during the phasic movements of RBD will be compared to the recordings obtained at the same level during a motor task.
  Other Names: Synchronised video-polysomnography and STN local field potentials recordings.

SUMMARY:
To compare the electrical activity of SubThalamic Nuclei (STN), by mean of local field potentials recordings, during the phasic behaviours of RBD with the electrical activity recorded at this level during the execution of voluntary movements during the "off" and the "on" phases in patients with RBD secondary to PD.

DETAILED DESCRIPTION:
Patient with severe Parkinson's disease (PD) with motor fluctuations are akinetic and bradykinetic during the "off" phases. Their motor status dramatically improves during "on" phases, due to the effect of dopaminergic agents.

In the off phases, the plasmatic levels of dopaminergic drugs are the lowest. The plasmatic levels of dopaminergic drugs are also very low during nocturnal sleep.

Nevertheless, PD patients may show vigorous and rapid movements during REM Behaviour Disorder (RBD). Thirty-three to 46% of the patients with PD have RBD.

Akinesia and bradykinesia are the consequence of a hyperactivity of the SubThalamic Nuclei (STN). The electrophysiological correlate of this hyperactivity causing akinesia and bradykinesia is represented by STN beta activity, recorded by local field potentials.

STN beta activity is not present during the execution of a voluntary movement at an "on" phase. Levodopa therapy, which can revert akinesia and bradykinesia, also suppress STN beta activity in PD patients The STN is the surgical target for Deep Brain Stimulation (DBS) of the basal ganglia to improve the motor symptoms of PD.

The STN has bilateral connections with the laterodorsal nucleus/pedunculopontine tegmentum (LDT/PPN), a key structure for REM sleep regulation.

The investigators hypothesize that during the execution of the phasic motor behaviours of RBD the pattern of discharge of STN differs from the one observed during voluntary movements in the "off" phase, in PD patients. In other terms, we expect the STN beta activity to disappear during the execution of phasic motor behaviors of RBD.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, 35 to 70 years old, with idiopathic PD (UKPDSBB criteria) with motor fluctuations
* having RBD according to the International Classification of Sleep Disorders, 2nd edition (ICSD-2) criteria
* Eligible to neurosurgical treatment of PD by implantation of intracranial electrodes for the DBS of STN
* Giving a written informed consent
* Affiliated to the French social security program

Exclusion Criteria:

* Atypical or secondary parkinsonian syndrome
* Cognitive impairment which may compromise the understanding and patient's participation to the protocol (Mattis dementia rating scale score ≥ 136)
* Patient under guardianship, trusteeship or judicial protection
* Pregnancy or breastfeeding
* Patient participating to another clinical research study in the same period

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-06; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
STN 8-30 Hz mean power | Outcome measure is assessed during the 2 nights and the two days following the implantation of the electrode in the STN.
  Difference of the mean power of the 8-30 Hz frequency band at the NST during the phasic movements of TCSP and during the execution voluntary movements in the "off" phase.

SECONDARY OUTCOMES:
Difference of the mean power of the 8-13 Hz, 14-30 Hz and 60-90 Hz frequency bands at the NST during the phasic movements of TCSP and during the execution voluntary movements in the "off" phase. | Outcome measures are assessed at days 2 and 3 and nights 1 and 2.
Difference of the mean power of the 8-30 Hz and 60-90 Hz frequency bands at the NST during the phasic movements of TCSP and during the execution voluntary movements in the "on" phase. | Outcome measures are assessed at days 2 and 3 and nights 1 and 2.
Frequency spectrum at NST REM sleep without atonia and REM sleep with atonia. | Outcome measures are assessed at days 2 and 3 and nights 1 and 2.
Frequency spectrum at the NST during non REM sleep (N1, N2 and N3 stages), REM sleep (R) and nocturnal wake. | Outcome measures are assessed at days 2 and 3 and nights 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Pietro-Luca RATTI, MD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - University Hospital of Purpan, Toulouse, Midi-Pyrénées
  - University Hospital of Rangueil, Toulouse, Midi-Pyrénées

REFERENCES:
- [Background] AASM (2005). International classification of sleep disorders, 2nd ed.: Diagnostic and coding manual. Westchester, IL, American Academy of Sleep Medicine.
- [Background] Benarroch EE. Subthalamic nucleus and its connections: Anatomic substrate for the network effects of deep brain stimulation. Neurology. 2008 May 20;70(21):1991-5. doi: 10.1212/01.wnl.0000313022.39329.65. No abstract available. PMID 18490619
- [Background] Boeve BF, Silber MH, Saper CB, Ferman TJ, Dickson DW, Parisi JE, Benarroch EE, Ahlskog JE, Smith GE, Caselli RC, Tippman-Peikert M, Olson EJ, Lin SC, Young T, Wszolek Z, Schenck CH, Mahowald MW, Castillo PR, Del Tredici K, Braak H. Pathophysiology of REM sleep behaviour disorder and relevance to neurodegenerative disease. Brain. 2007 Nov;130(Pt 11):2770-88. doi: 10.1093/brain/awm056. Epub 2007 Apr 5. PMID 17412731
- [Background] Brown P, Williams D. Basal ganglia local field potential activity: character and functional significance in the human. Clin Neurophysiol. 2005 Nov;116(11):2510-9. doi: 10.1016/j.clinph.2005.05.009. Epub 2005 Jul 18. PMID 16029963
- [Background] Buot, A., M. L. Welter, et al. (2012).
- [Background] Cassidy M, Mazzone P, Oliviero A, Insola A, Tonali P, Di Lazzaro V, Brown P. Movement-related changes in synchronization in the human basal ganglia. Brain. 2002 Jun;125(Pt 6):1235-46. doi: 10.1093/brain/awf135. PMID 12023312
- [Background] De Cock VC, Vidailhet M, Leu S, Texeira A, Apartis E, Elbaz A, Roze E, Willer JC, Derenne JP, Agid Y, Arnulf I. Restoration of normal motor control in Parkinson's disease during REM sleep. Brain. 2007 Feb;130(Pt 2):450-6. doi: 10.1093/brain/awl363. PMID 17235126
- [Background] Drouin, N., L. Allard, et al. (2011). Sleep staging using Subdermal Wire Electrodes during intracerebral EEG recordings (abstract 1.133). American Epilepsy Society 65th annual meeting. Baltimore, MD., U.S.A.
- [Background] Fernandez-Mendoza J, Lozano B, Seijo F, Santamarta-Liebana E, Ramos-Platon MJ, Vela-Bueno A, Fernandez-Gonzalez F. Evidence of subthalamic PGO-like waves during REM sleep in humans: a deep brain polysomnographic study. Sleep. 2009 Sep;32(9):1117-26. doi: 10.1093/sleep/32.9.1117. PMID 19750916
- [Background] Fumagalli, M., G. Giannicola, et al. (2011).
- [Background] Hammond C, Bergman H, Brown P. Pathological synchronization in Parkinson's disease: networks, models and treatments. Trends Neurosci. 2007 Jul;30(7):357-64. doi: 10.1016/j.tins.2007.05.004. Epub 2007 May 25. PMID 17532060
- [Background] Hsu, Y. T., H. Y. Lai, et al. (2012).
- [Background] Iber, C., S. Ancoli-Israel, et al. (2007). The AASM Manual for the Scoring of Sleep and Associated Events. Rules, Terminology and Technical Specifications. Westchester, IL, American Academy of Sleep Medicine.
- [Background] Kuhn AA, Trottenberg T, Kivi A, Kupsch A, Schneider GH, Brown P. The relationship between local field potential and neuronal discharge in the subthalamic nucleus of patients with Parkinson's disease. Exp Neurol. 2005 Jul;194(1):212-20. doi: 10.1016/j.expneurol.2005.02.010. PMID 15899258
- [Background] Levy R, Ashby P, Hutchison WD, Lang AE, Lozano AM, Dostrovsky JO. Dependence of subthalamic nucleus oscillations on movement and dopamine in Parkinson's disease. Brain. 2002 Jun;125(Pt 6):1196-209. doi: 10.1093/brain/awf128. PMID 12023310
- [Background] Luppi, P. H., O. Clement, et al. (2011).
- [Background] Marceglia S, Fumagalli M, Priori A. What neurophysiological recordings tell us about cognitive and behavioral functions of the human subthalamic nucleus. Expert Rev Neurother. 2011 Jan;11(1):139-49. doi: 10.1586/ern.10.184. PMID 21158561
- [Background] Martinez-Martin, P., C. Rodriguez-Blazquez, et al. (2013).
- [Background] Mena-Segovia J, Bolam JP, Magill PJ. Pedunculopontine nucleus and basal ganglia: distant relatives or part of the same family? Trends Neurosci. 2004 Oct;27(10):585-8. doi: 10.1016/j.tins.2004.07.009. PMID 15374668
- [Background] Nishida, N., T. Murakami, et al. (2011).
- [Background] Oudiette, D., S. Leu-Semenescu, et al. (2012).
- [Background] Rivlin-Etzion M, Marmor O, Heimer G, Raz A, Nini A, Bergman H. Basal ganglia oscillations and pathophysiology of movement disorders. Curr Opin Neurobiol. 2006 Dec;16(6):629-37. doi: 10.1016/j.conb.2006.10.002. Epub 2006 Nov 3. PMID 17084615
- [Background] Rodriguez-Oroz, M. C., J. Lopez-Azcarate, et al. (2011).
- [Background] Sixel-Döring, F., E. Trautmann, et al. (2011).
- [Background] Stefani A, Galati S, Peppe A, Bassi A, Pierantozzi M, Hainsworth AH, Bernardi G, Orlacchio A, Stanzione P, Mazzone P. Spontaneous sleep modulates the firing pattern of parkinsonian subthalamic nucleus. Exp Brain Res. 2006 Jan;168(1-2):277-80. doi: 10.1007/s00221-005-0175-y. Epub 2005 Nov 18. PMID 16328297
- [Background] Trenkwalder, C., R. Kohnen, et al. (2011).
- [Background] Urbain N, Gervasoni D, Souliere F, Lobo L, Rentero N, Windels F, Astier B, Savasta M, Fort P, Renaud B, Luppi PH, Chouvet G. Unrelated course of subthalamic nucleus and globus pallidus neuronal activities across vigilance states in the rat. Eur J Neurosci. 2000 Sep;12(9):3361-74. doi: 10.1046/j.1460-9568.2000.00199.x. PMID 10998119
- [Background] Urrestarazu E, Iriarte J, Alegre M, Clavero P, Rodriguez-Oroz MC, Guridi J, Obeso JA, Artieda J. Beta activity in the subthalamic nucleus during sleep in patients with Parkinson's disease. Mov Disord. 2009 Jan 30;24(2):254-60. doi: 10.1002/mds.22351. PMID 18951542
- [Background] Visser, M., J. Marinus, et al. (2004).
- [Background] Weinberger M, Mahant N, Hutchison WD, Lozano AM, Moro E, Hodaie M, Lang AE, Dostrovsky JO. Beta oscillatory activity in the subthalamic nucleus and its relation to dopaminergic response in Parkinson's disease. J Neurophysiol. 2006 Dec;96(6):3248-56. doi: 10.1152/jn.00697.2006. Epub 2006 Sep 27. PMID 17005611
- [Background] Williams D, Kuhn A, Kupsch A, Tijssen M, van Bruggen G, Speelman H, Hotton G, Loukas C, Brown P. The relationship between oscillatory activity and motor reaction time in the parkinsonian subthalamic nucleus. Eur J Neurosci. 2005 Jan;21(1):249-58. doi: 10.1111/j.1460-9568.2004.03817.x. PMID 15654862